CLINICAL TRIAL: NCT06856304
Title: Percutaneous Internal Ring Suturing Versus Conventional Laparoscopic Repair of Congenital Inguinal Hernia: a Prospective Randomized Study
Brief Title: Percutaneous Internal Ring Suturing Versus Conventional Laparoscopic Repair of Congenital Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0107373
Record Dates: First submitted 2025-02-25; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2022-09

CONDITIONS: Pediatrics; Inguinal Hernia Repair
Keywords: Laparoscopy; inguinal hernia; PIRS; sac disconnection; Narrowing of the internal ring
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): laparoscopic disconnection of the hernia sac and narrowing of the internal ring
  Interventions: Procedure: laparoscopic disconnection of the hernia sac
- Group B (Experimental): Percautaneous internal ring suturing
  Interventions: Procedure: Percutaneous internal ring suturing

INTERVENTIONS:
Procedure: laparoscopic disconnection of the hernia sac — disconnection of the hernial sac at the level of the internal ring using hook diathermy with sweeping the vas and the vessels away till completely separating them from the edges of the sac, then narrowing of the internal ring by appling a vicryl 3/0 suture between the ilipubic tract and the transverse arch of the transversus abdominus muscle
  Arms: Group A
Procedure: Percutaneous internal ring suturing — A single umbilical trocar was placed through a supraumbilical incision, and then the surgeon stood on the same side of the hernia. To choose the location for the needle puncture, the position of the IIR was assessed by pressing the inguinal region from the outside with the tip of a forceps. Under laparoscopic-guided vision, the previously prepared 18-gauge injection needle threaded with the monofilament suture was introduced into the abdominal wall through a skin puncture at the lateral edge of the internal ring. With the movements of the tip of the needle, the thread passed under the peritoneum, over the lateral half of the IIR. The thread was pushed through the barrel of the needle into the abdominal cavity and eventually made a loop. The needle was pulled out, leaving the loop of the thread inside the abdomen by hanging the loop on the endoscope this prevented the extraction of the loop with the needle and thus prevented repeating this step. Next, the thread loop was pulled out of t
  Arms: Group B

SUMMARY:
Background:comparison between percutaneous internal ring suturing vs Conventional Laparoscopic Repair of Congenital Inguinal Hernia in male patients. Methods : this is a prospective randomized study including 109 male patients with 120 CIHs Patients were randomly categorized into two groups. Group A were subjected to laparoscopic disconnection of the hernia sac and narrowing of the internal ring (IR). Group B underwent PIRS. The intended primary outcome was recurrence within 1 year, besides comparing the two techniques regarding operative time, efficacy, safety, cosmetic outcome, and postoperative complications.

DETAILED DESCRIPTION:
Introduction Since the 1990s laparoscopy has gained popularity in the management of Congenital inguinal hernia (CIH). Several laparoscopic techniques have been described, including laparoscopic disconnection of the hernial sac with narrowing of the internal ring (IIR) which was described to mimic the open technique, and the extraperitoneal approach involves using various types of needles under laparoscopic guidance to percutaneously secure a suture circumferentially around the internal ring, thus obliterating the sac opening. This study compared the short-term outcome of percutaneous internal ring suturing (PIRS) versus laparoscopic disconnection of the hernial sac with narrowing of the internal ring in children.

Materials and Methods: This study included 109 male patients with 120 CIHs during the period from May 2022 to May 2024. Patients were randomly categorized into two groups. Group A were subjected to laparoscopic disconnection of the hernia sac and narrowing of the internal ring (IR). Group B underwent PIRS. The intended primary outcome was recurrence within 1 year, besides comparing the two techniques regarding operative time, efficacy, safety, cosmetic outcome, and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* male patients
* age of 6 month to 5years
* reduciable congenital inguinal hernia either unilateral or bilateral.

Exclusion Criteria:

* incarcerated CIH
* recurrent CIH
* patients with undescended testis,
* patients with hydrocele,
* patients with chronic comorbidity such as congenital heart disease and severe chest troubles

Ages: 6 Months to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — only male patients were included
Enrollment: 109 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
operative time | the time estimated during the operation
  time of the procedure estimated after trocars insertion and Inflation of the abdomen till deflation of the abdomen
intraoperative safety | the time estimated during the operation
  injury of the vas deffernce , spermatic vessels , bleeding
Recurrence of the inguinal hernia | 1 year
  postoperative swelling in the inguinal region with gurgling sensation

SECONDARY OUTCOMES:
cosmesis | 1 year
  postoperative scar

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abouheba, Assistant Professor, Study Director — University of Alexandria
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No